CLINICAL TRIAL: NCT03361657
Title: Arterial to End-Tidal Carbon Dioxide Difference During Pediatric Laparoscopic Surgeries
Acronym: PaCO2-EtCO2
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, principal investigator, Assiut University
Other Study IDs: 17300081
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Intraoperative Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One sample: Laparoscopic surgeries will be performed according to the standard surgical and anesthesia protocols. Pneumo-peritoneum will be achieved using non-heated non-humidified CO2 with the intra-abdominal pressure (IAP) maintained at 10-12mmHg

SUMMARY:
Studying the arterial to end-tidal carbon dioxide difference in children undergoing laparoscopic surgeries under different intra-abdominal pressures is of extreme importance. This is because both hyper and hypocarbia are detrimental in this vulnerable age group.

DETAILED DESCRIPTION:
Capnography provides a non-invasive estimate of arterial CO2 levels and allows clinicians to modify mechanical ventilation settings in order to maintain normocapnia. Normally, a positive gap between arterial CO2 and ETCO2 of approximately 0.5 kPa is assumed in a healthy patient and ventilation settings are adjusted accordingly. However, the correlation between PaCO2 and PetCO2 during laparoscopic surgery is inconsistent mainly due to inter- and intra-individual variability. Discrepancies between arterial carbon dioxide and End-tidal carbon dioxide measures have been demonstrated in ventilated children with cyanotic congenital heart disease , infants with respiratory failure and during visceral and urological laparoscopic surgery. Moreover, as the increase in PaCO2 is directly proportional to the level of intra-abdominal pressure (IAP) used, variations in the arterial to end-tidal carbon dioxide difference can be also expected with different levels of IAP used.

ELIGIBILITY:
Inclusion Criteria:

* Children with the following inclusion criteria;
* Weight: 10-30 kg.
* Age: 1-6 years.
* Sex: both males and females.
* ASA physical status: I, II.
* Operation: elective laparoscopic surgeries that last more than 45 min.

Exclusion Criteria:

Patients will be excluded if they have;

* Patients with any perioperative cardiovascular or respiratory event occurred which made the study intervention clinically unacceptable,
* Patients with unsatisfactory preoperative peripheral arterial oxygen saturation,
* Patients with unsatisfactory preoperative hemoglobin level, neurological or psychiatric disease,
* Children with a BMI >95th percentile for age.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children scheduled for laparoscopic surgery of Weight: 10-30 kg, Age: 1-6 years, both males and females,ASA physical status: I, II.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Correlation between the Arterial to end-tidal carbon dioxide | Intraoperative
  The arterial CO2 will be analysed from the blood gas and the endtidal carbon dioxide will be recorded from the capnography tracing.

SECONDARY OUTCOMES:
PaCO2-ETCO2 Difference | Intraoperative
  The arterial CO2 will be analysed from the blood gas and the endtidal carbon dioxide will be recorded from capnography.
Heart rate | Intraoperative
  The heart rate will be continuously monitored, intraoperatively
The noninvasive systolic and diastolic arterial blood pressure | intraoperative
  The non invasive systolic and diastolic arterial blood pressure will be recorded at fixed intervals

CONTACTS AND LOCATIONS:
Overall Officials: Hala Abdelghaffar, MD, Principal Investigator — professor in Anesthesia department, faculty of medicine, Assiut university, Assiut, Egypt
Locations (1):
- Assiut university Pediatric hospital, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdel-Ghaffar HS, Bakr MA, Osman MA, Hanna SGL, Ali WN. End-tidal carbon dioxide measurements as a surrogate to arterial carbon dioxide during pediatric laparoscopic surgeries: a prospective observational cohort study. Braz J Anesthesiol. 2024 Sep-Oct;74(5):744261. doi: 10.1016/j.bjane.2021.07.036. Epub 2021 Aug 16. PMID 34411630